CLINICAL TRIAL: NCT02698371
Title: NCCL Direct Composite Restoration Performance With Self-Etch and Multimode Adhesives Clinical Trial
Brief Title: NCCL Direct Composite Restoration Performance With Self-Etch and Multimode Adhesives
Acronym: SEMMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Patrícia Manarte Monteiro, Associate Professor, University Fernando Pessoa
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: FCS-UFP-2014-04-2015-07-19; EC/011/2015 (Other: INFARMED)
Record Dates: First submitted 2016-02-03; First posted 2016-03-03 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Dental Adhesives/Restorations Performance
Keywords: composite resins; dental restoration; adhesives; non-carious cervical lesions; clinical effectiveness; Adhese universal; Futurabond U; Futurabond DC; self-etch; multimode/universal; clinical trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- FBDC-SE (G1; Control) (Active Comparator): Futurabond DC (single dose blister) will be applied as thickness to the enamel/dentine and rub into the tooth surface for 20s; FBDC drying layer for at least 5s with an air syringe; This adhesive layer will be light-cured with a light emitting diode unit (LED light), with an intensity of 1000mW/cm2, during 20s.
  Interventions: Device: G1-Control: Futurabond®DC-SE (FBDC_SE)
- FBDC-SE-EE (G2; Control ) (Active Comparator): Etch with 36% phosphoric acid, during 30s in enamel structures. Remove the 36% phosphoric acid with water during 1 minute. The remove of water excess will be done with weak air spray, not to dry the dentine completely. The dentine surface must slightly remain wet. Application of Futurabond DC (FBDC) as self-etch mode simultaneously in dentin and enamel, and the light-cured (LED light; 1000mW/cm2), during 20s.
  Interventions: Device: G2-Control: Futurabond®DC_SE_EE
- FBU-ER (G3) (Other): FuturabondU® (FBU) apply in enamel and dentin as etch-and-rinse (ER) mode. Etching of the dental hard tissue phosphoric acid (15s in dentin and 30s in enamel) and then rinse with water for 1 min. Dry off excess moisture with a gentle stream of air. Activating FBU SingleDose. FBU adhesive will be homogeneously applied to all cavity surfaces and rub in for 20s using the Single Tim; This adhesive layer will be light-cured with a light emitting diode unit, with an intensity of 1000mW/cm2 during 20s.
  Interventions: Device: G3: Futurabond® U - ER (FBU_ER)
- FBU-SE (G4) (Other): FuturabondU® (FBU) apply in enamel and dentin as SE mode. Activating FBU SingleDose. FBU adhesive will be homogeneously apply to all cavity surfaces and rub in for 20 s using the Single Tim; Dry off the adhesive layer with dry, oil-free air for at least 5 s in order to remove any solvents. This adhesive layer will be light-cured with a light emitting diode unit (LED light), with an intensity of 1000mW/cm2, during 20 seconds.
  Interventions: Device: G4: Futurabond® U - SE (FBU_SE)
- ADU-ER (G5) (Other): Adhese®Universal (ADU) apply by etch-and-rinse (ER) mode. Etching of the dental hard tissue phosphoric acid (15 seconds in dentin and 30 seconds in enamel); Etch agent rinse with water for 1 minute. Dry off excess moisture with a gentle stream of air. Keep dentin dry, do not over dry; Adhesive ADU will be scrubbed into the tooth surface (enamel and dentin) for at least 20 seconds. Adhesive will be dispersed with compressed air until a glossy, immobile film layer results.Light-curing for 10 s with a light emitting diode unit (LED light), with an intensity of 1000mW/cm2 for 20s.
  Interventions: Device: G5: Adhese® Universal - ER (ADU_ER)
- ADU-SE (G6) (Other): Adhese®Universal (ADU)apply by self-etch (SE) mode. Starting with the enamel, thoroughly coat the tooth surfaces (enamel and dentin) to be treated with ADU; Adhesive will be scrubbed into the tooth surface for at least 20 seconds. Adhesive will be dispersed with compressed air until a glossy, immobile film layer results.Light-curing for 20 s with a light emitting diode unit (LED light), with an intensity of 1000mW/cm2.
  Interventions: Device: G6: Adhese® Universal - SE (ADU_SE)

INTERVENTIONS:
Device: G1-Control: Futurabond®DC-SE (FBDC_SE) — Futurabond®DC (FBDC) adhesive by self-etch (SE) mode bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Futurabond®DC_Self-etch mode (FBDC_SE)
  Arms: FBDC-SE (G1; Control)
Device: G2-Control: Futurabond®DC_SE_EE — Futurabond®DC adhesive by self-etch mode with selective enamel etching (FBDC-SE-EE) bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Futurabond®DC_selective Enamel Etching (FBDC_SE_EE)
  Arms: FBDC-SE-EE (G2; Control )
Device: G3: Futurabond® U - ER (FBU_ER) — FuturabondU® (FBU) adhesive by etch-and-rinse (ER) mode, bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Futurabond® U_Etch-and-Rinse mode (FBU_ER)
  Arms: FBU-ER (G3)
Device: G4: Futurabond® U - SE (FBU_SE) — FuturabondU® (FBU) adhesive by self-etch (SE) mode, bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Futurabond® U - Self-Etch mode (FBU_SE)
  Arms: FBU-SE (G4)
Device: G5: Adhese® Universal - ER (ADU_ER) — Adhese®Universal (ADU) adhesive by etch-and-rinse (ER) mode, bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Adhese® Universal - Etch-and-rinse mode (ADU_ER)
  Arms: ADU-ER (G5)
Device: G6: Adhese® Universal - SE (ADU_SE) — Adhese®Universal (ADU) adhesive by self-etch (SE) mode, bonding in NCCls restorations, was randomly assigned to premolar or molar teeth ensuring that this adhesive/mode is only apllied once in each participant.
  Other Names: Adhese® Universal - Self-Etch mode (ADU_SE)
  Arms: ADU-SE (G6)

SUMMARY:
The purpose is to evaluate/compare clinical effectiveness of dual cure (DC) all-in-one Self-Etch (Futurabond® DC (FBDC)) adhesive and multimode/universal (Futurabond® U (FU) and Adhese® Universal (AU)) adhesives, with or without selective enamel etching, in non-carious cervical lesions (NCCL), during 24th months, using Word Dental Federation (FDI) and United States Public Health Services (USPHS) criteria.

The null hypotheses are:

H0 - Bonding to NCCLs with DC-SE and SE-Universal adhesives with SE strategies will result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance in a period of 24th month evaluation; H0 - Bonding to NCCLs with DC-SE and SE-Universal adhesives with SE strategies will result in similar restorations (aesthetic, functional and biologic) success rates over 24th month evaluation; H0 - Bonding to NCCLs with DC-SE and SE-Universal adhesives with SE strategies will result in similar restoration retention rates in a period of 24th month evaluation; H0 - Bonding to NCCLs DC-SE with enamel pre-etching and Universal adhesives with ER adhesive strategy will result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance in a period of 24thmonth evaluation; H0 - Bonding to NCCLs DC-SE with enamel pre-etching and Universal adhesives with ER adhesive strategy will result in similar restorations (aesthetic, functional and biologic) success rates over 24th month evaluation; H0 - Bonding to NCCLs DC-SE with enamel pre-etching and Universal adhesives with ER adhesive strategy will result in similar restoration retention rates in a period of 24th month evaluation; H0 - Bonding to NCCLs with FBDC or FU (DC adhesives) and AU (Light-curing adhesive) with SE or ER adhesive strategies will result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance in a period of 24th month evaluation; H0 - Bonding to NCCLs with FBDC or FU (DC adhesives) and AU (Light-curing adhesive) with SE or ER adhesive strategies will result in similar restorations (aesthetic, functional and biologic) success rates over 24th month evaluation; H0 - Bonding to NCCLs with FBDC or FU (DC adhesives) and AU (Light-curing adhesive) with SE or ER adhesive strategies will result in similar restoration retention rates in a period of 24th month evaluation; H0 - FDI or USPHS criteria evaluation outcomes not differ for the same data.

DETAILED DESCRIPTION:
2.1- DESIGN The trial design will follow the Consolidated Standards of Reporting Trials (CONSORT) statement (1, 2).

Prospective, double blind clinical trial; randomized allocation of NCCL restorations by six adhesion treatment groups (6 arms: G1 to G6) for examination of restorations performance. Study will take place in University Fernando Pessoa - Faculty of Health Sciences (UFP-FHS), Dental Medicine School Clinic. Participants recruitment estimated between November 2015 and April 2016.

The study is scheduled to last 24th months. Baseline clinical observation will be done 30 days after placement of adhesion restoration (First data), second observation at 12 months and last evaluation at 24 months (Data for Statistical analysis). Clinical trial may continue for similar assessment intervals, after 24th months evaluation. This situation requires new analysis according to clinical and economics conditions, at that time.

2.2- POPULATION AND PARTICIPANT SELECTION

All participants will be informed (Written and verbal information) about the trial conditions and purposes, but will not be aware of what tooth will received the adhesion treatment. Written informed consent, according to World Medical Association Declaration of Helsinki (3), will be obtained from all participants prior to starting the treatment. University Fernando Pessoa Ethics Committee review and approved the present protocol. This clinical trial is done according to the National Law 21/2014, of 16 April, and was analysed, approved and authorized by the National Competent Authorities:

* INFARMED, National Authority of Medicines and Health Products, IP (No.EC/011/2015; DPS/DM/450.10.053/2015/0314; Authorization at 4th August 2015)
* CEIC, National Ethics Committee for Clinical Research (No.20150305; Approved at 3th August 2015)
* CNPD, Portuguese Data Protection Authority (Authorization and registry 6430/2015 at 7 July 2015; No.2536/2015).

The decision to participate in this study is voluntary as well as the decision to refuse participation and decision of withdrawal of the same, at any time of the study course, are rights of the patient/participant. The operator (Dentist and Associate Professor of FHS-UFP) inform the patient/participant in all aspects related to the study. Refusal of patient participation, the participant's withdrawal and revocation of consent to participate in this study are rights of the patient/participant without any consequences or reprisal, and without interference in the relationship between users and teachers/ researchers / University, clinical entities.

SAMPLE:

Patients with clinical diagnosis of non-carious cervical lesion (NCCLs) located in pre-molars/molars (PM/M) teeth, with cavity dimensions defined in the study design.

Two hundred and ten restorations will be performed, randomized in order to be allocated to six interventions (G1 to G6 arms), named as adhesion intervention groups.

Within this trial, the number of teeth to be restored by participant will be between a minimum of 1 and a maximum of 6. The allocation of the study group (G1 to G6) to a particular tooth is random with the information available to the operator/principal investigator in sealed envelopes and previously prepared by the investigator-professional statistics. The allocation of the study group (G1, G2, G3, G4, G5, G6) to each tooth for a patient is performed randomly, but ensuring that the distribution of the groups is not repeated in the same patient. For this purpose, 210 envelopes with 35 sequences of 6 study groups will be organized by the statistical investigator (wherein each order of 6 groups is randomized).

2.3- STUDY ADHESION ARMS Six groups (G1 to G6) of NCCL restorations will be randomized allocated according to adhesion strategy intervention.

2.4- OPERATOR / EXAMINERS CALIBRATION Operator will do one restoration of each group in order to identify all steps involved in the application technique. This procedure will be done three times, with one week, interval. All restorations done by the same calibrated operator. Three experienced and calibrated dentists, not involved with the restoring procedures and therefore blinded to the group assignment, will perform the clinical evaluation. For training purposes, the examiners observed 10 photographs that were representative of each score for each criterion, in 10 cervical restorations (not included in this trial), each one, on two consecutive days. An intra-examiner and inter-examiner agreement will be calculated.

Medical Devices Composition (According to Manufactures, Voco and Ivoclar Vivadent Safety data sheets for Adhesives and products):

1. Futurabond® DC (Voco, Cuxhaven, Germany) Batch No.1532592:

   Liquid 1. Acidic adhesive monomer; BIS-GMA (5-10%), 2-HEMA (5-10%); pH-value 1.5 Liquid 2. Ethanol (50-100%); Initiator (2.5-5%) Mixture. organic acids, BIS-GMA, 2-HEMA, TMPTMA, campherchinon, amines (DABE), BHT, catalysts, fluorides and ethanol.
2. Futurabond® U (Voco, Cuxhaven, Germany) Batch No.1543141:

   Liquid 1. 2-hidroxyethyl methacrylate (2-HEMA) (25-50%); BIS-GMA (25-50%); HEDMA (10-25%); Acidic adhesive monomer (5-10%); Urethanedimethacrylate (UDMA) (5-10%); catalysts (≤ 2.5%); pH-value 2.3 Liquid 2. Ethanol (50-100%); Initiator (2.5-5%); catalysts (≤ 2.5%)
3. Ivoclar Vivadent's Adhese® Universal (Ivoclar Vivadent AG, Liechtenstein) Batch No.U35131:

   Composition/information on ingredients; mixture of substances Liquid: 2-hydroxyethyl methacrylate (20-<25%); bisphenol A diglycidyl ether dimethacrylate (20-<25%); ethanol (10-<25%); decamethylene dimethacrylate (3-<10%); Methacrylated phosphoric acid ester (3-<10%); campherquinone (1-<2.5%); 2-dimethylaminoethyl methacrylate (1-<2.5%); 2,6-di-tert-butyl-p-cresol (0.1-<0.3%). (MDP-Methacryloyloxydecyl dihydrogen phosphate; MCAP- Methecrylated carboxylic acid polymer; HEMA-Hydroxyethil methacrylate; Bis-GMA_ Bisphenol A glycidyl methacrylate; D3MA- Decandiol dimethacrylate); pH-value 2.5-3.0.
4. Vococid® (Voco, Cuxhaven, Germany) Batch No.152135: 35% orthophosphoric acid; 2.5- DATA REGISTRY/PROTECTION AND RESTORATIONS PROCEDURES Only in the registration database (with access to the principal investigator and other team members, with the exception of the statistical investigator for the purposes of observational clinical records) there should be registration/membership of this key with the code-process of patients. The database in question will be lodged in own servers with restricted access levels and well identified. The servers that lodge the photos/ records and the database belong to Dental School Clinic of Faculty of Health Sciences - UFP and are located in data centre with fully controlled access. This mechanism ensures the concealment of identity of the user in records file, having access to them only the investigator and research team (except investigator of statistics). This mechanism fulfilled the recommendation and Authorisation of CNPD, Portuguese Data Protection Authority (Authorization and registry 6430/2015 at 7 July 2015; Case 2536/2015).

Appointment and restorative procedures, in accordance with the following steps:

One week, before the Restorative procedure (1st appointment): Inform the patient (Written/Verbal); Patient signature of informed consent; Fulfilment of the project clinical file (patient identification, general clinical summary, oral clinic examination, oral hygiene state); Dental prophylaxis with fluoride toothpaste and water with a nylon brush. Vitality tests (cold and hot) executed with spray Endo cool (ethyl chloride) and warm instrument; Pre-operative sensitivity evaluation by applying air for 10 seconds from a dental syringe placed 2 cm from the tooth surface (4); NCCLs cavities will be evaluated according to the degree (1, 2, 3, 4) of sclerotic dentin (5), cavity dimensions (H-height, W-width, and D-depth) in millimetres (mm) and geometry (evaluated by profile photograph, as Angles Acute (A), Severe (S), Obtuse (O) (4); 1st Appointment-Intervention: Initial intra-oral/cavity surface and tooth digital photography; Teeth anaesthesia with 3% mepivacaine (Scandinibsa, Sintra Business Park, Portugal); Operatory field isolation with cotton rolls and retraction floss (Ultradent). All cavities cleaned with pumice and water in a rubber cup, followed by rinsing and drying. Selection composite colour by shade guide; Adhesive interventions according to G1 to G6 arms assignment. Adhesive systems will be used as SingleDose mode. Composite restorations (AdmiraFusion Universal nano-hybrid composite) with incremental filling technique (two increments maximum), light-cured (LED Unit) with an intensity of 1000mW/cm2, during 40 seconds. Restorations will be finished immediately with diamond disks (OptiDisc® medium 40μm; Kerr) and burns. Polishing performed with diamond-impregnated silicone polishers (Dimanto, Voco, CuxHaven) during 10 seconds. Intra-oral digital photography of the restoration.

2.6- CLINICAL FOLLOW-UP Baseline (30 days after restoration), 12th (NCCLs observation) and 24th months (for statistical analysis) Appointments

1 - Intra-oral digital photography of the NCCL restoration; 2- Post-operative sensitivity evaluation by applying air for 10 seconds from a dental syringe placed 2 cm from the tooth surface (4); 3 - Direct evaluation by 3 calibrated examiners according to FDI (6, 7) and USPHS (8); 4- Data register Study variable definition - Clinical/direct observation and performance evaluation acceptance by means of FDI and USPHS criteria.

2.7- DATA BASE AND STATISTICAL ANALISYS Data statistical analysis and description according to aims of this trial; Specific program for statistical data analysis (IBM(c) SPSS(c) Statistics vs. 23 or later) will be used. Differences will be considered to be significant at p<0.05.

2.8- OBSERVATIONS REGARDING SAMPLE CALCULATION Was assumed that the minimum number of bonded restorations to be held in each of the six arms (G1 to G6) is 35 (210 restorations). The researchers did not have detailed information that allows the estimation of the sample size based on power analysis (the effect of the expected difference to the end of the time considered for the study). Thus, using rules of thumb usually considered in research situations where there is no prior information concerning the performance evaluation of these class IIa medical devices available on the market. In this case, considering that it intends to make a prospective longitudinal study, to determine factors associated with failure rate and reduced clinical performance (effect) criteria of the restorations, and to detect effects depends the number of events (failure, for example, or other event that is to be considered in the defined evaluation criteria) and not the number of participants, the thumb rules stipulate a minimum of 10 cases by group. Moreover, when considering an "simple" analysis comparison using a McNemar test (repeated measures) in six groups would be necessary in total, including at least 80 cases (to restore teeth) in the sample. When considering at least 35 restorations by group, researchers are greatly increasing the minimum number stipulated in any of the aforementioned techniques. In addition, clinical studies previously performed on this issue (between 2004 and 2012) relative to the post-market clinical evaluation performance of class IIa medical devices, in the context of restorative dentistry field, has enabled to measure a minimum of 30 restorations as viable for determining events in a short/medium-term as the clinical performance evaluation of a similar nature of medical devices.

2.9- GOOD CLINICAL PRACTICE FOR CLINICAL RESEARCH Reporting mechanism of possible adverse incident during the investigation will be held according to Medical Devices (MD) commercially available in the market, so it interprets and assumes the issue as applicable to assumptions in the Portuguese National Law (Article 22) 21/2014, of 16 April, calling up a mechanism for reporting any incidents inherent to medical devices or resulting from the use of medical devices. In this way, and considering the type of intervention to carry out in this research (restoration of very small extension of NCCL with dental adhesives), the medical devices (Adhesive systems) are not described in the literature and not known records for the occurrence of undesirable incidents, with interpretative effects as Serious or Unexpected "adverse incidents". However, and according to good clinical practice for clinical research, the reporting mechanism of Serious or Unexpected incidents (protocol version FHS-UFP-FFP-2014 April-19.07.2015) for this research are approved by CEIC (National Ethics Committee for Clinical Research (No.20150305; Approved at 3th August 2015).

Sponsor reports annually to CEIC and INFARMED a list of all suspected serious adverse events, during this period as well as a report on the safety of participants, if applicable. Under the study protocol (Version FCS-UFP-FFP-2014 April-19.07.2015), all the possible non-serious adverse events such as, clinical signs or symptoms associated with loss of aesthetic, functional and biological performance of restorations and situations described in the instructions, labelling and safety data sheets of medical devices or even, without incident and security maintenance data of the participants the sponsor notifies the CEIC and INFARMED, only by the final evaluation of this study (two years of clinical performance), as set forth in article 24th of Law 21/2014 of 16 April, which will include a report of suspicious occurrences and safety records and, if applicable, in the clinical trial in the period Evaluation of two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* ages up to 18 years old and less than 65 years old
* Patients with diagnosis and treatment required of dental structure loss in cervical vestibular surfaces with non-bacterial or chemical origin, which is non-carious cervical lesions (NCCL) in premolar/molar teeth (These lesions have to be non-carious, non-retentive, deeper than 1 mm, and involve both the enamel and dentin of vital teeth without mobility. The cavo-surface margin cannot involve more that 50% of enamel.)

Exclusion Criteria:

* Patients with a number of teeth inferior than 20 in occlusion;
* If the tooth is not vital;
* Chronic periodontal disease;
* Incapacity to return to follow-up;
* To participate in another clinical evaluation in course at that time;
* Medical, psychiatric history or pharmacotherapy to compromise the protocol
* Pregnancy;
* Allergies and idiosyncratic answers to the ingredients of the products;
* Fixed orthodontic treatment;
* Teeth support for fixed prosthodontic treatments;
* Teeth or structures of support with pulpa injury in transition phase;
* Periodontal surgery in the 3 previous months;
* Severe bruxism;
* Extremely poor oral hygiene;
* Patient refuse to voluntary participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Manarte-Monteiro, PhD, Principal Investigator — University Fernando Pessoa
Locations (1):
- University Fernando Pessoa, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645
- [Background] Ritter AV, Heymann HO, Swift EJ Jr, Sturdevant JR, Wilder AD Jr. Clinical evaluation of an all-in-one adhesive in non-carious cervical lesions with different degrees of dentin sclerosis. Oper Dent. 2008 Jul-Aug;33(4):370-8. doi: 10.2341/07-128. PMID 18666493
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Science Committee Project 2/98--FDI World Dental Federation study design (Part I) and criteria for evaluation (Part II) of direct and indirect restorations including onlays and partial crowns. J Adhes Dent. 2007;9 Suppl 1:121-47. PMID 18341239
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Derived] Manarte-Monteiro P, Domingues J, Teixeira L, Gavinha S, Manso MC. Multi-Mode adhesives performance and success/retention rates in NCCLs restorations: randomised clinical trial one-year report. Biomater Investig Dent. 2019 Nov 6;6(1):43-53. doi: 10.1080/26415275.2019.1684199. eCollection 2019. PMID 31998871
- See also: University Fernando Pessoa — http://international.ufp.pt/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Dental School Clinic of the Faculty of Health Sciences - UFP.
Pre-assignment Details: 54 participants were screened. Of those, 38 participants met inclusion criteria and were enrolled.
Units Other Than Participants: NCCLs restorations
Groups:
- All Participants: Each participant is enrolled in several randomly allocated arms/groups (G1, G2, G3, G4, G5, G6) and received one to six NCCLs restorations in Premolar/molar teeth.
Period: All Participants Flow
Arm/Group | All Participants
Started (Baseline) | 38; 210 NCCLs restorations
Completed (Two years recall) | 35; 193 NCCLs restorations
Not Completed | 3; 17 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: FBDC-SE (G1; Control) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with FBDC-SE (G1control Arm/Group).)
Completed (Two years recall) | 32; 32 NCCLs restorations
Not Completed | 3; 3 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: FBDC-SE-EE (G2; Control ) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with FBDC-SE-EE (G2 control Arm/group))
Completed (Two years recall) | 32; 32 NCCLs restorations
Not Completed | 3; 3 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: FBU-ER (G3) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with FBU-ER (G3 Arm/group))
Completed (Two years recall) | 32; 32 NCCLs restorations
Not Completed | 3; 3 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: FBU-SE (G4) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with FBU-SE (G4 Arm/group))
Completed (Two years recall) | 32; 32 NCCLs restorations
Not Completed | 3; 3 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: ADU-ER (G5) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with ADU-ER (G5 Arm/group))
Completed (Two years recall) | 32; 32 NCCLs restorations
Not Completed | 3; 3 NCCLs restorations
Not completed — Lost to Follow-up | 3
Period: ADU-SE (G6) Arm/Group Flow
Arm/Group | All Participants
Started (Baseline) | 35; 35 NCCLs restorations (Each participant received one NCCLs restoration with ADU-SE (G6 Arm/group))
Completed (Two years recall) | 33; 33 NCCLs restorations
Not Completed | 2; 2 NCCLs restorations
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Each participant is enrolled in several Arms/Groups and received 1 to 6 NCCLs restorations; The allocation of the arm/group (G1, G2, G3, G4, G5, G6) to each NCCLs of each participant was performed ensuring that the distribution of the arms/groups was not repeated in the same participant.
Units Other Than Participants: NCCLs restorations
Arm/Group | All Participants
Number analyzed (Participants) | 38
Number analyzed (NCCLs restorations) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] — NCCLs restorations per arm/group distribution, according to the participant mean age. Population: Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  years
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control group) Arm/Group | 50.8 (10.9)
    FBDC-SE-EE (G2; Control group) Arm/Group | 51.4 (10.1)
    FBU-ER (G3) Arm/Group | 50.6 (10.4)
    FBU-SE (G4) Arm/Group | 51.5 (9.8)
    ADU-ER (G5) Arm/Group | 50.5 (11.1)
    ADU-SE (G6) Arm/Group | 50.8 (10.8)
Sex: Female, Male [Count of Units; unit: NCCLs restorations] — Population: NCCLs restorations per arm/group distribution, according to the participant sex
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: Female | 15
    FBDC-SE (G1; Control Group) Arm/Group: Male | 20
    FBDC-SE-EE (G2; Control Group) Arm/Group: Female | 16
    FBDC-SE-EE (G2; Control Group) Arm/Group: Male | 19
    FBU-ER (G3) Arm/Group: Female | 16
    FBU-ER (G3) Arm/Group: Male | 19
    FBU-SE (G4) Arm/Group: Female | 16
    FBU-SE (G4) Arm/Group: Male | 19
    ADU-ER (G5) Arm/Group: Female | 14
    ADU-ER (G5) Arm/Group: Male | 21
    ADU-SE (G6) Arm/Group: Female | 14
    ADU-SE (G6) Arm/Group: Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Systemic pathologies at baseline [Count of Units; unit: NCCLs restorations] — Population: NCCLs restorations per arm/group distribution, according to the participant systemic pathologies (yes/no) at baseline. Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: No | 16
    FBDC-SE (G1; Control Group) Arm/Group: yes | 19
    FBDC-SE-EE (G2; Control group) Arm/Group: No | 14
    FBDC-SE-EE (G2; Control group) Arm/Group: yes | 21
    FBU-ER (G3) Arm/Group: No | 15
    FBU-ER (G3) Arm/Group: yes | 20
    FBU-SE (G4) Arm/Group: No | 14
    FBU-SE (G4) Arm/Group: yes | 21
    ADU-ER (G5) Arm/Group: No | 16
    ADU-ER (G5) Arm/Group: yes | 19
    ADU-SE (G6) Arm/Group: No | 16
    ADU-SE (G6) Arm/Group: yes | 19
Oral hygiene at baseline [Count of Units; unit: NCCLs restorations] — Population: NCCLs restorations per arm/group distribution, according to the participant oral hygiene (very good/good) at baseline. Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: Very good | 23
    FBDC-SE (G1; Control Group) Arm/Group: Good | 12
    FBDC-SE-EE (G2; Control group) Arm/Group: Very good | 25
    FBDC-SE-EE (G2; Control group) Arm/Group: Good | 10
    FBU-ER (G3) Arm/Group: Very good | 25
    FBU-ER (G3) Arm/Group: Good | 10
    FBU-SE (G4) Arm/Group: Very good | 24
    FBU-SE (G4) Arm/Group: Good | 11
    ADU-ER (G5) Arm/Group: Very good | 23
    ADU-ER (G5) Arm/Group: Good | 12
    ADU-SE (G6) Arm/Group: Very good | 22
    ADU-SE (G6) Arm/Group: Good | 13
Smoking habits at baseline [Count of Units; unit: NCCLs restorations] — Population: NCCLs restorations per arm/group distribution, according to the participant smoking habits (yes/no) at baseline. Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: No | 30
    FBDC-SE (G1; Control Group) Arm/Group: Yes | 5
    FBDC-SE-EE (G2; Control group) Arm/Group: No | 30
    FBDC-SE-EE (G2; Control group) Arm/Group: Yes | 5
    FBU-ER (G3) Arm/Group: No | 30
    FBU-ER (G3) Arm/Group: Yes | 5
    FBU-SE (G4) Arm/Group: No | 30
    FBU-SE (G4) Arm/Group: Yes | 5
    ADU-ER (G5) Arm/Group: No | 29
    ADU-ER (G5) Arm/Group: Yes | 6
    ADU-SE (G6) Arm/Group: No | 30
    ADU-SE (G6) Arm/Group: Yes | 5
Daily cigarettes (NCCLs restorations in smoker participants) at baseline [Mean (Standard Deviation); unit: cigarettes per day] — Population: NCCLs restorations per arm/group distribution, according to the participant Daily cigarettes (NCCLs restorations in smoker participants) at baseline. Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  cigarettes per day
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group | 2.1 (5.6)
    FBDC-SE-EE (G2; Control group) Arm/Group | 1.6 (4.7)
    FBU-ER (G3) Arm/Group | 1.6 (4.7)
    FBU-SE (G4) Arm/Group | 1.6 (4.7)
    ADU-ER (G5) Arm/Group | 2.2 (5.6)
    ADU-SE (G6) Arm/Group | 1.8 (5.3)
NCCLs Tooth Type [Count of Units; unit: NCCLs restorations] — Population: Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: Pre-molar tooth | 29
    FBDC-SE (G1; Control Group) Arm/Group: Molar tooth | 6
    FBDC-SE-EE (G2; Control group) Arm/Group: Pre-molar tooth | 32
    FBDC-SE-EE (G2; Control group) Arm/Group: Molar tooth | 3
    FBU-ER (G3) Arm/Group: Pre-molar tooth | 32
    FBU-ER (G3) Arm/Group: Molar tooth | 3
    FBU-SE (G4) Arm/Group: Pre-molar tooth | 27
    FBU-SE (G4) Arm/Group: Molar tooth | 8
    ADU-ER (G5) Arm/Group: Pre-molar tooth | 30
    ADU-ER (G5) Arm/Group: Molar tooth | 5
    ADU-SE (G6) Arm/Group: Pre-molar tooth | 26
    ADU-SE (G6) Arm/Group: Molar tooth | 9
NCCLs Sclerotic Dentin Degree [Count of Units; unit: NCCLs restorations] — Degree 1= No sclerosis present. Dentine is light yellow or whitish in colour with little discoloration; Dentine is opaque, with little translucency or transparency. Degree 2= More than category 1, but less than 50% of the difference between categories 1 and 4. Degree 3= Less than category 4, but more than 50% of the difference between categories 1 and 4. Degree 4= Significant sclerosis present. Dentine is dark yellow or even discoloured (brownish). Dentine appears glassy, with significant translucency or transparency evident. Population: Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: Degree 1 | 29
    FBDC-SE (G1; Control Group) Arm/Group: Degree 2 | 4
    FBDC-SE (G1; Control Group) Arm/Group: Degree 3 | 0
    FBDC-SE (G1; Control Group) Arm/Group: Degree 4 | 2
    FBDC-SE-EE (G2; Control group) Arm/Group: Degree 1 | 24
    FBDC-SE-EE (G2; Control group) Arm/Group: Degree 2 | 7
    FBDC-SE-EE (G2; Control group) Arm/Group: Degree 3 | 1
    FBDC-SE-EE (G2; Control group) Arm/Group: Degree 4 | 3
    FBU-ER (G3) Arm/Group: Degree 1 | 26
    FBU-ER (G3) Arm/Group: Degree 2 | 5
    FBU-ER (G3) Arm/Group: Degree 3 | 0
    FBU-ER (G3) Arm/Group: Degree 4 | 4
    FBU-SE (G4) Arm/Group: Degree 1 | 20
    FBU-SE (G4) Arm/Group: Degree 2 | 7
    FBU-SE (G4) Arm/Group: Degree 3 | 3
    FBU-SE (G4) Arm/Group: Degree 4 | 5
    ADU-ER (G5) Arm/Group: Degree 1 | 23
    ADU-ER (G5) Arm/Group: Degree 2 | 5
    ADU-ER (G5) Arm/Group: Degree 3 | 4
    ADU-ER (G5) Arm/Group: Degree 4 | 3
    ADU-SE (G6) Arm/Group: Degree 1 | 24
    ADU-SE (G6) Arm/Group: Degree 2 | 7
    ADU-SE (G6) Arm/Group: Degree 3 | 0
    ADU-SE (G6) Arm/Group: Degree 4 | 4
NCCls Cavity Geometry (Internal angle shape, degree º) [Count of Units; unit: NCCLs restorations] — Population: Each participant is enrolled in several arms and received 1 to 6 NCCLs restorations.
  NCCLs restorations
    number analyzed (Participants) | 35
    number analyzed (NCCLs restorations) | 35
    FBDC-SE (G1; Control Group) Arm/Group: Acute (<45º) | 13
    FBDC-SE (G1; Control Group) Arm/Group: Acute-to-Right (45º- 90º) | 9
    FBDC-SE (G1; Control Group) Arm/Group: Obtuse (>90º) | 13
    FBDC-SE-EE (G2; Control group) Arm/Group: Acute (<45º) | 17
    FBDC-SE-EE (G2; Control group) Arm/Group: Acute-to-Right (45º- 90º) | 11
    FBDC-SE-EE (G2; Control group) Arm/Group: Obtuse (>90º) | 7
    FBU-ER (G3) Arm/Group: Acute (<45º) | 14
    FBU-ER (G3) Arm/Group: Acute-to-Right (45º- 90º) | 11
    FBU-ER (G3) Arm/Group: Obtuse (>90º) | 10
    FBU-SE (G4) Arm/Group: Acute (<45º) | 14
    FBU-SE (G4) Arm/Group: Acute-to-Right (45º- 90º) | 9
    FBU-SE (G4) Arm/Group: Obtuse (>90º) | 12
    ADU-ER (G5) Arm/Group: Acute (<45º) | 15
    ADU-ER (G5) Arm/Group: Acute-to-Right (45º- 90º) | 8
    ADU-ER (G5) Arm/Group: Obtuse (>90º) | 12
    ADU-SE (G6) Arm/Group: Acute (<45º) | 11
    ADU-SE (G6) Arm/Group: Acute-to-Right (45º- 90º) | 12
    ADU-SE (G6) Arm/Group: Obtuse (>90º) | 12

OUTCOME MEASURES:

1. Primary Outcome: Esthetic, Functional and Biological Clinical Performance Adhesive/Adhesion Mode of NCCLs Restoration, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Clinical Performance Acceptance was expressed as the number of NCCls restorations scored as "1-Clinically excellent/ very good", "2-Clinically good (after correction, very good)", "3-Clinically sufficient/ satisfactory (minor shortcomings with no adverse effects but not adjustable without damage to the tooth)", "4-Clinically unsatisfactory (repair for prophylactic reasons)". NCCls restorations with not acceptable performance were scored as "5-Clinically poor (replacement necessary)" for clinical properties. NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Groups:
- FBDC-SE (G1; Control Group): Futurabond®DC (FBDC) adhesive by self-etch (SE) mode in NCCls cavities randomly assigned to premolar or molar teeth: FBDC rubbered in enamel and dentine for 20s, then dryed for at least 5s with an air syringe and then light-cured.
- FBDC-SE-EE (G2; Control Group): FBDC adhesive by self-etch mode with selective enamel etching (FBDC-SE-EE) in NCCls cavities randomly assigned to premolar or molar teeth: Enamel etched with 36% phosphoric acid for 30s and then removed with water during 1 minute; finally, FBDC applied by SE mode, simultaneously in dentin and enamel and light-cured.
- FBU-ER (G3): FuturabondU® (FBU) adhesive by etch-and-rinse (ER) mode in NCCls cavities randomly assigned to premolar or molar teeth: Etching of dental tissues with 36% phosphoric acid (15s in dentin and 30s in enamel) and then rinse with water for 1 min; Dryed off the excess moisture with a gentle stream of air. FBU rubbered in enamel and dentine for 20s, then dyed for at least 5s and then light-cured.
- FBU-SE (G4): FBU adhesive by self-etch (SE) mode in NCCls cavities randomly assigned to premolar or molar teeth: FBU rubbered in enamel and dentine for 20s, then dyed for at least 5s and then, light-cured.
- ADU-ER (G5): Adhese®Universal (ADU) adhesive by etch-and-rinse (ER) mode in NCCls cavities randomly assigned to premolar or molar teeth: Etching of dental tissues with 36% phosphoric acid (15s in dentin and 30s in enamel) and then rinse with water for 1 min; Dryed off the excess moisture with a gentle stream of air. ADU scrubbled in enamel and dentine for 20s, then dyed for at least 5s and then light-cured.
- ADU-SE (G6): ADU adhesive by self-etch (SE) mode in NCCLs cavities randomly assigned to premolar or molar teeth: ADU scrubbled in enamel and dentine for 20s, then dyed for at least 5s and then light-cured.
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Esthetic-FDI- 24 Month: Acceptance Performance | 29 | 30 | 29 | 30 | 32 | 33
  Esthetic-FDI- 24 Month: Not Acceptance Performance | 0 | 0 | 0 | 0 | 0 | 0
  Esthetic-FDI- 24 Month: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  Functional-FDI- 24 Month: Acceptance Performance | 29 | 30 | 29 | 30 | 32 | 33
  Functional-FDI- 24 Month: Not Acceptance Performance | 3 | 2 | 3 | 2 | 0 | 0
  Functional-FDI- 24 Month: NCCLs restorations missing | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-FDI-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-FDI-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-FDI-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-FDI-24 Month (included in Functional Not Acceptance Performance count of Units) | 0 | 0
  Biological-FDI- 24 Month: Acceptance Performance | 29 | 30 | 29 | 30 | 32 | 33
  Biological-FDI- 24 Month: Not Acceptance Performance | 0 | 0 | 0 | 0 | 0 | 0
  Biological-FDI- 24 Month: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance between baseline and 24 month follow-up;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.025, McNemar
Statistical Analysis 2: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC-SE (G1) and MM-SE(G4G6) result in similar restorations (aesthetic, functional and biologic) success rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.189, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC-SE (G1) and MM-SE (G4G6) adhesives result in similar restoration retention rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.189, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance from baseline to 24 month follow-up;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.025, McNemar
Statistical Analysis 5: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC-SE-EE (G2) and MM-ER (G3G5) result in similar restorations (aesthetic, functional and biologic) success rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.747, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC-SE-EE (G2) and MM-ER (G3G5) result in similar restoration retention rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.747, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis
Statistical Analysis 8: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4) and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar restorations (aesthetic, functional and biologic) success rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis — Applied for rows/Categories- Acceptance Vs Not Acceptance Functional-FDI comparison between G1G2 and G3G4 and G5G6 Arms success rate from baseline to 24 month recall. For Esthetic and Biological-FDI comparison p values were > 0.05. Adjusted P-values
Statistical Analysis 9: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4) and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar restoration retention rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis — Applied for rows/Categories- Acceptance Vs Not Acceptance Retention-FDI comparison between G1G2 and G3G4 and G5G6 Arms retention rate from baseline to 24 month recall. Adjusted P-values

2. Primary Outcome: Esthetic, Functional and Biological Clinical Performance Adhesive/Adhesion Mode of NCCLs Restoration, Graded on a 4-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Clinical Performance Acceptance was expressed as the number of NCCls restorations scored as "Alfa" and "Bravo". NCCls restorations with not acceptable performance were scored as "Charlie" for Esthetic properties, for Retention criteria and for Biological properties, and also scored "Delta" for Marginal Adaptation criteria. NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Groups:
- FBU-SE (G4): FBU adhesive by self-etch (SE) mode in NCCls cavities randomly assigned to premolar or molar teeth: FBU rubbered in enamel and dentine for 20s, then dyed for at least 5s and then light-cured.
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Esthetic-USPHS- 24 Month: Acceptance Performance | 29 | 30 | 29 | 30 | 32 | 33
  Esthetic-USPHS- 24 Month: Not Acceptance Performance | 0 | 0 | 0 | 0 | 0 | 0
  Esthetic-USPHS- 24 Month: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  Functional-USPHS- 24 Month: Acceptance Performance | 29 | 30 | 29 | 30 | 32 | 33
  Functional-USPHS- 24 Month: Not Acceptance Performance | 3 | 2 | 3 | 2 | 0 | 0
  Functional-USPHS- 24 Month: NCCLs restorations missing | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-USPHS-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-USPHS-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-USPHS-24 Month (included in Functional Not Acceptance Performance count of Units) | NA — NCCLs restorations missing due to retention lost were classified as Not Acceptance Performance for Functional-USPHS-24 Month (included in Functional Not Acceptance Performance count of Units) | 0 | 0
  Biological-USPHS- 24 Month: Acceptance Performance | 28 | 28 | 28 | 27 | 30 | 32
  Biological-USPHS- 24 Month: Not Acceptance Performance | 1 | 2 | 1 | 3 | 2 | 1
  Biological-USPHS- 24 Month: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.025, McNemar
Statistical Analysis 2: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.189, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC-SE (G1) and MM-SE (G4G6) adhesives result in similar restoration retention rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.189, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) clinical (aesthetic, functional and biologic) behaviour/performance;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.025, McNemar
Statistical Analysis 5: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); [analysis description as in outcome 1, analysis 5]; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.154, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC-SE-EE (G2) and MM-ER (G3G5) result in similar restoration retention rates;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.747, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); [analysis description as in outcome 1, analysis 7]; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis
Statistical Analysis 8: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); [analysis description as in outcome 1, analysis 8]; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis
Statistical Analysis 9: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); [analysis description as in outcome 1, analysis 9]; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.070, Kruskal-Wallis

3. Primary Outcome: FDI or USPHS Criteria Evaluation Outcomes for Esthetic, Functional and Biological Parameters, at 24th Month Follow-up.
Description: FDI or USPHS criteria evaluation outcomes for Esthetic, Functional and Biological parameters, at 24th month follow-up were expressed as the number os NCCLs With Clinical Acceptance for each parameter. NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Esthetic, Functional and Biological parameters, using FDI and USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Groups:
- FBDC-SE-EE (G2; Control Group): FBDC adhesive by self-etch mode with selective enamel etching (FBDC-SE-EE) in NCCls cavities randomly assigned to premolar or molar teeth: Enamel etched with 36% phosphoric acid for 30s and then removed with water during 1 minute; finally, FBDC applied by SE mode, simultaneously in dentin and enamel, and light-cured.
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  FDI-Esthetic: NCCLs restorations Acceptable | 29 | 30 | 29 | 30 | 32 | 33
  FDI-Esthetic: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  FDI-Esthetic: NCCLs restorations Not Acceptable | 0 | 0 | 0 | 0 | 0 | 0
  USPHS-Esthetic: NCCLs restorations Acceptable | 29 | 30 | 29 | 30 | 32 | 33
  USPHS-Esthetic: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  USPHS-Esthetic: NCCLs restorations Not Acceptable | 0 | 0 | 0 | 0 | 0 | 0
  FDI-Functional: NCCLs restorations Acceptable | 29 | 30 | 29 | 30 | 32 | 33
  FDI-Functional: NCCLs restorations missing | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for FDI-Functional category (included in NCCLs restorations FDI-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for FDI-Functional category (included in NCCLs restorations FDI-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for FDI-Functional category (included in NCCLs restorations FDI-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for FDI-Functional category (included in NCCLs restorations FDI-Functional Count of Units) | 0 | 0
  FDI-Functional: NCCLs restorations Not Acceptable | 3 | 2 | 3 | 2 | 0 | 0
  USPHS-Functional: NCCLs restorations Acceptable | 29 | 30 | 29 | 30 | 32 | 33
  USPHS-Functional: NCCLs restorations missing | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for USPHS-Functional category (included in NCCLs restorations USPHS-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for USPHS-Functional category (included in NCCLs restorations USPHS-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for USPHS-Functional category (included in NCCLs restorations USPHS-Functional Count of Units) | NA — NCCLs restorations not observed due to retention/marginal integrity lost were scored as Not Acceptable for USPHS-Functional category (included in NCCLs restorations USPHS-Functional Count of Units) | 0 | 0
  USPHS-Functional: NCCLs restorations Not Acceptable | 3 | 2 | 3 | 2 | 0 | 0
  FDI-Biological: NCCLs restorations Acceptable | 29 | 30 | 29 | 30 | 32 | 33
  FDI-Biological: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  FDI-Biological: NCCLs restorations Not Acceptable | 0 | 0 | 0 | 0 | 0 | 0
  USPHS-Biological: NCCLs restorations Acceptable | 28 | 28 | 28 | 27 | 30 | 32
  USPHS-Biological: NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
  USPHS-Biological: NCCLs restorations Not Acceptable | 1 | 2 | 1 | 3 | 2 | 1
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0: FDI or USPHS criteria Esthetic outcomes not differ at 24th month follow-up regarding Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4) and ADU (G5G6) adhesive, with SE or SE-ER/ER modes; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Chi-squared — Applied for rows/Categories- Acceptance Vs Not Acceptance Esthetic of FDI and of USPHS comparison; Applied to G1G2; G3G4 and G5G6 separately
Statistical Analysis 2: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0: FDI or USPHS criteria Functional outcomes not differ at 24th month follow-up regarding Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4) and ADU (G5G6) adhesive, with SE or SE-ER/ER modes; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Chi-squared — Applied for rows/Categories- Acceptance Vs Not Acceptance Functional of FDI and of USPHS comparison; Applied to G1G2; G3G4 and G5G6 separately
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0: FDI or USPHS criteria Biological outcomes not differ at 24th month follow-up regarding Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4) and ADU (G5G6) adhesive, with SE or SE-ER/ER modes; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.998, Chi-squared — Applied for rows/Categories- Acceptance Vs Not Acceptance Biologic FDI and of USPHS comparison; Applied to G1G2; G3G4 and G5G6 separately

4. Secondary Outcome: Surface Luster, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Surface Luster Clinical Acceptance was expressed as the number of NCCls restorations classified as "(11)-Luster comparable to enamel", "(12)-Slightly dull, not noticeable from speaking distance", "(13)-Dull surface but acceptable if covered with film of saliva", "(14)- Rough surface, cannot be masked by saliva film, simple polishing is not sufficient. Further intervention necessary". NCCls restorations with not acceptable Surface Luster were classified as "(15)-Quite rough, unacceptable plaque retentive surface". NCCLs restorations not observed due to retention lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Surface Luster, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score (11) | 28 | 30 | 29 | 30 | 32 | 32
  Score (12) | 1 | 0 | 0 | 0 | 0 | 1
  Score (13) | 0 | 0 | 0 | 0 | 0 | 0
  Score (14) | 0 | 0 | 0 | 0 | 0 | 0
  Score (15) | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Surface Luster Performance at 24 Month Follow-up recall; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.029, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) Surface Luster-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Surface Luster performance at 24 Month Follow-up recall;; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.002, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) Surface Luster-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Surface Luster performance at 24 Month Follow-up recall; Test type: Equivalence — alpha value of 0.05 was considered; p = 0.618, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) Surface Luster-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

5. Secondary Outcome: Staining Margin, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Staining Margin Clinical Acceptance was expressed as the number of NCCls restorations classified as "(21)-No surface staining", "(22)-Minor staining, easily removable", "(23)-Moderate surface staining, also present on other teeth, not aesthetically unacceptable", "(24)-Surface staining present on the restoration and is unacceptable; major intervention necessary for improvement". NCCls restorations with not acceptable Staining Margin were classified as "(25)-Severe staining and/or subsurface staining (generalized or localized); not accessible for intervention". NCCLs restorations not observed due to retention lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Staining Margin, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 21 | 26 | 29 | 28 | 28 | 30 | 30
  Score 22 | 3 | 0 | 0 | 1 | 0 | 1
  Score 23 | 0 | 1 | 1 | 1 | 1 | 2
  Score 24 | 0 | 0 | 0 | 0 | 1 | 0
  Score 25 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Staining Margin Performance at 24 Month Follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.009, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) Staining Margin-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Staining Margin Performance at 24 Month Follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.059, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) Staining Margin-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Staining Margin performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.829, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) Staining Margin-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

6. Secondary Outcome: Colour Stability and Translucency, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Colour Stability and Translucency Clinical Acceptance was expressed as the number of NCCls restorations classified as "(31)-Good colour match no difference in shade and translucency", "(32)-Minor deviations", "(33)-Clear deviation but acceptable. Does not affect aesthetics", "(34)-(Localised) clinically unsatisfactory but can be corrected by repair". NCCls restorations with not acceptable Colour Stability and Translucency were classified as "(35)-Unacceptable. Replacement necessary". NCCLs restorations not observed due to retention lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Colour Stability and Translucency, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 31 | 29 | 30 | 29 | 30 | 30 | 32
  Score 32 | 0 | 0 | 0 | 0 | 2 | 1
  Score 33 | 0 | 0 | 0 | 0 | 0 | 0
  Score 34 | 0 | 0 | 0 | 0 | 0 | 0
  Score 35 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Colour Stability performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p < 0.001, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) Colour Stability-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Colour Stability performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p < 0.001, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Colour Stability-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Colour Stability performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.064, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Colour Stability-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

7. Secondary Outcome: Fractures and Retention, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Fractures and Retention Clinical Acceptance was expressed as the number of NCCls restorations classified as "(41)-Restoration retained, no fractures/cracks", "(42)-Small hairline crack", "(43)-Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity or proximal contact", "(44)-Chipping fractures which damage marginal quality or proximal contacts; bulk fractures with or without partial loss(less than half of the restoration)". NCCls restorations with not acceptable Fractures and Retention were classified "(45)-Partial or complete loss of restoration".
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Fractures and Retention, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 41 | 29 | 29 | 29 | 27 | 32 | 32
  Score 42 | 0 | 0 | 0 | 2 | 0 | 1
  Score 43 | 0 | 0 | 0 | 0 | 0 | 0
  Score 44 | 0 | 1 | 0 | 1 | 0 | 0
  Score 45 | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Fractures and Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.006, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Fractures and Retention-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Fractures and Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.020, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Fractures and Retention-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Fractures and Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.054, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Fractures and Retention-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

8. Secondary Outcome: Marginal Adaptation, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Marginal Adaptation Clinical Acceptance was expressed as the number of NCCls restorations classified as "(51)-Harmonious outline, no gaps, no discoloration", "(52)-Marginal gap (50 µm) or Small marginal fracture removable by polishing", "(53)-Gap< 150 µm not removable or Severe small enamel or dentin fractures", "(54)- Gap> 250 µm or dentine exposed or Chip fracture damaging margins or Notable enamel or dentine wall fracture", "(55)-Filling is loose but in situ". NCCLs restorations not observed due to retention lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Marginal Adaptation, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 51 | 21 | 29 | 24 | 24 | 27 | 27
  Score 52 | 5 | 0 | 3 | 3 | 3 | 2
  Score 53 | 3 | 1 | 2 | 3 | 2 | 4
  Score 54 | 0 | 0 | 0 | 0 | 0 | 0
  Score 55 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Marginal Adaptation performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.010, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Marginal Adaptation-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Marginal Adaptation performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.071, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Marginal Adaptation-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Marginal Adaptation performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.898, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Marginal Adaptation-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

9. Secondary Outcome: Postoperative Hypersensibility, Tooth Vitality, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Postoperative Hypersensibility, Tooth Vitality Clinical Acceptance was expressed as the number of NCCls restorations classified as "(61)-No hypersensitivity, normal vitality", "(62)-Low hypersensitivity for a limited period of time, normal vitality", "(63)-Premature/slightly more intense or Delayed/weak sensitivity; no subjective complaints, no treatment needed", "(64)-Premature/very intense or Extremely delayed/weak with subjective complaints or Negative sensitivity intervention necessary but not replacement". NCCls restorations with not acceptable Postoperative Hypersensibility, Tooth Vitality criteria were classified as (65)-Very intense, acute pulpitis or no vital; Endodontic treatment is necessary and restoration has to be replaced".NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Postoperative Hypersensibility, Tooth Vitality, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 61 | 29 | 28 | 29 | 28 | 30 | 32
  Score 62 | 0 | 2 | 0 | 2 | 2 | 1
  Score 63 | 0 | 0 | 0 | 0 | 0 | 0
  Score 64 | 0 | 0 | 0 | 0 | 0 | 0
  Score 65 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Postoperative Hypersensibility, Tooth Vitality performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.317, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Postoperative Hypersensibility, Tooth Vitality-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Postoperative Hypersensibility, Tooth Vitality performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.180, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Postoperative Hypersensibility, Tooth Vitality-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Postoperative Hypersensibility, Tooth Vitality performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.918, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Postoperative Hypersensibility, Tooth Vitality-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

10. Secondary Outcome: Recurrence of Caries, Erosion, Abfraction, Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Recurrence of Caries, Erosion, Abfraction Clinical Acceptance was expressed as the number of NCCls restorations classified as "(71)-No secondary or primary caries", "(72)-Very small and localized. No operative treatment required", "(73)-Larger areas of: Demineralisation or Erosion or Abrasion/abfraction in dentine, localized and accessible and can be repaired", "(74)-Caries with cavitation or Erosion in dentine or Abrasion/abfraction in dentine Localized and accessible and can be repaired". NCCls restorations with not acceptable Recurrence of Caries, Erosion, Abfraction criteria were classified as "(75)-Deep secondary caries or exposed dentine that is not accessible for repair of restoration". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Recurrence of Caries, Erosion, Abfraction, using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 71 | 29 | 29 | 29 | 29 | 32 | 33
  Score 72 | 0 | 0 | 0 | 1 | 0 | 0
  Score 73 | 0 | 0 | 0 | 0 | 0 | 0
  Score 74 | 0 | 1 | 0 | 0 | 0 | 0
  Score 75 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Recurrence of Caries, Erosion, Abfraction performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.317, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Recurrence of Caries, Erosion, Abfraction-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Recurrence of Caries, Erosion, Abfraction performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = .317, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Recurrence of Caries, Erosion, Abfraction-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Recurrence of Caries, Erosion, Abfraction performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.575, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Recurrence of Caries, Erosion & Abfraction-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

11. Secondary Outcome: Tooth Integrity (Enamel Cracks), Graded on a 5-point Scale, Using FDI Criteria at 24 Month Follow-up Recall
Description: Tooth Integrity (enamel cracks) Clinical Acceptance was expressed as the number of NCCls restorations classified as "(81)-Complete integrity", "(82)-Small margin enamel(<150 µm) or Hairline crack in enamel (<150 µm not probable)", "(83)-Enamel split(<250 µm) or Crack< 250 µm, no adverse effects", "(84)-Major enamel split (gap>250 µm or dentine or base exposed) or Crack>250 µm (probe penetrates)". NCCls restorations with not acceptable Tooth Integrity (enamel cracks) criteria were classified as "(85)-Cusp or tooth fracture". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Tooth Integrity (enamel cracks), using FDI criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Score 81 | 26 | 30 | 27 | 26 | 28 | 32
  Score 82 | 3 | 0 | 2 | 3 | 3 | 1
  Score 83 | 0 | 0 | 0 | 1 | 1 | 0
  Score 84 | 0 | 0 | 0 | 0 | 0 | 0
  Score 85 | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Tooth Integrity (enamel cracks) performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.020, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Tooth Integrity (enamel cracks)-FDI comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Tooth Integrity (enamel cracks) performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.107, Wilcoxon (Mann-Whitney) — Applied for all rows/Categories (graded on a 5-point scale) of Tooth Integrity (enamel cracks)-FDI comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Tooth Integrity (enamel cracks) performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.592, Kruskal-Wallis — Applied for all rows/Categories (graded on a 5-point scale) of Tooth Integrity (enamel cracks)-FDI comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

12. Secondary Outcome: Surface Staining, Graded on a 3-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Surface Staining Clinical Acceptance was expressed as the number of NCCls restorations classified as "(Alfa)- No staining in the restoration and/or the tooth" or "(Bravo)-Slight staining in the restoration and/or the tooth". NCCls restorations with not acceptable Surface Staining were classified as "(Charlie)-The staining penetrated in the restoration and/or the tooth in a pulpal direction". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Surface Staining, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Alfa | 29 | 30 | 29 | 30 | 32 | 33
  Bravo | 0 | 0 | 0 | 0 | 0 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Surface Staining performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Surface Staining-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Surface Staining performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Surface Staining-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Surface Staining performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Kruskal-Wallis — Applied for rows/categories alfa/bravo/charlie of Surface Staining-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

13. Secondary Outcome: Marginal Discoloration, Graded on a 3-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Marginal Discoloration Clinical Acceptance was expressed as the number of NCCls restorations classified as "(Alfa)-No discoloration along the margin between the restoration and adjacent tooth" or "(Bravo)-Slight discoloration along the margin between the restoration and the adjacent tooth (removable, usually localized)". NCCls restorations with not acceptable Marginal Discoloration were classified as "(Charlie)-Deep staining cannot be polished away". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Marginal Discoloration, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Alfa | 25 | 28 | 27 | 27 | 29 | 31
  Bravo | 4 | 2 | 2 | 3 | 3 | 2
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Marginal Discoloration performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.011, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Marginal Discoloration-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Marginal Discoloration performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.034, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Marginal Discoloration-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Marginal Discoloration performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.885, Kruskal-Wallis — Applied for rows/categories alfa/bravo/charlie of Marginal Discoloration-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

14. Secondary Outcome: Color Match, Graded on a 3-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Color Match Clinical Acceptance was expressed as the number of NCCls restorations classified as "(Alfa)-Restoration matches the adjacent tooth structure in color and translucency" or "(Bravo)-Light mismatch in color, shade or translucency between the restoration and the adjacent tooth". NCCls restorations with not acceptable Color Match were classified as "(Charlie)-The mismatch in color and translucency is outside the acceptable range of tooth color and translucency". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Color Match, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Alfa | 29 | 30 | 29 | 30 | 31 | 33
  Bravo | 0 | 0 | 0 | 0 | 1 | 0
  Charlie | 0 | 0 | 0 | 0 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Color Match performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 1.000, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Color Match-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Color Match performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.317, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Color Match-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Color Match performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.403, Kruskal-Wallis — Applied for rows/categories alfa/bravo/charlie of Color Match-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

15. Secondary Outcome: Retention, Graded on a 3-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Retention Clinical Acceptance was expressed as the number of NCCls restorations classified as "(Alfa)-Retained" or "(Bravo)-Partially retained". NCCls restorations with not acceptable Retention were classified as "(Charlie)-Missing".
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Retention, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Alfa | 29 | 29 | 29 | 29 | 32 | 33
  Bravo | 0 | 1 | 0 | 1 | 0 | 0
  Charlie | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.020, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Retention-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.020, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie of Retention-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Retention performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.040, Kruskal-Wallis — Applied for rows/categories alfa/bravo/charlie of Retention-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

16. Secondary Outcome: Marginal Integrity, Graded on a 4-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Marginal Integrity Clinical Acceptance was expressed as the number of NCCls restorations classified as "(Alfa)-No visible evidence of crevice along the margin", "(Bravo)-Visible evidence of a crevice along the margin into which the explorer will penetrate"or "(Charlie)-Dentin or the base is exposed". NCCls restorations with not acceptable Marginal Integrity were classified as "(Delta)-Restoration is fractured, mobile or missing".
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Marginal Integrity, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  Alfa | 23 | 28 | 24 | 24 | 27 | 29
  Bravo | 6 | 2 | 5 | 5 | 5 | 4
  Charlie | 0 | 0 | 0 | 1 | 0 | 0
  Delta | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Marginal Integrity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p < 0.001, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie/delta of Marginal Integrity-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Marginal Integrity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p < 0.001, Wilcoxon (Mann-Whitney) — Applied for rows/categories alfa/bravo/charlie/delta of Marginal Integrity-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Marginal Integrity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.211, Kruskal-Wallis — Applied for rows/categories alfa/bravo/charlie/delta of Marginal Integrity-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

17. Secondary Outcome: Postoperative Sensitivity, Graded on a 2-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Postoperative Sensitivity Clinical Acceptance was expressed as the number of NCCls restorations classified as "(A)-No evidence of postoperative sensitivity". NCCls restorations with not acceptable Postoperative Sensitivity were classified as "(B)-Experience of postoperative sensitivity. NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Postoperative Sensitivity, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  (A)-No evidence | 28 | 28 | 29 | 27 | 30 | 32
  (B)-Experience | 1 | 2 | 0 | 3 | 2 | 1
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Postoperative Sensitivity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.102, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Postoperative Sensitivity-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Postoperative Sensitivity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.180, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Postoperative Sensitivity-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Postoperative Sensitivity performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.990, Kruskal-Wallis — Applied for rows/categories No Evidence vs Evidence of Postoperative Sensitivity-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

18. Secondary Outcome: Secondary Caries, Graded on a 2-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Secondary Caries Clinical Acceptance was expressed as the number of NCCls restorations classified as "(A)-No evidence of caries". NCCls restorations with not acceptable Secondary Caries criteria were classified as "(B)-Evidence of caries along the margin of the restoration. NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Secondary Caries, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  (A)-No evidence | 29 | 29 | 29 | 28 | 32 | 33
  (B)-Evidence | 0 | 1 | 0 | 2 | 0 | 0
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Secondary Caries performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.157, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Secondary Caries-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Secondary Caries performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.317, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Secondary Caries-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Secondary Caries performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.334, Kruskal-Wallis — Applied for rows/categories No Evidence vs Evidence of Secondary Caries-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

19. Secondary Outcome: Gingival Bleeding, Graded on a 2-point Scale, Using USPHS Criteria at 24 Month Follow-up Recall
Description: Gingival Bleeding Clinical Acceptance was expressed as the number of NCCls restorations classified as "(A)-No evidence of gingival bleeding adjacent to Class II restoration". NCCls restorations with not acceptable Gingival Bleeding criteria were classified as "(B)-Evidence of gingival bleeding adjacent to Class II restoration". NCCLs restorations not observed due to retention/marginal integrity lost were scored as "missing" for other categories.
Time Frame: 24 months
Population: Per protocol analysis Population, defined as participants completing (each one enrolled in several arms and received 1 to 6 restorations), and NCCLs restorations observed for Gingival Bleeding, using USPHS criteria, at 24 month recall.
Measure: Count of Units; unit: NCCLs restorations
Units Other Than Participants: NCCLs restorations
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 33
Number analyzed (NCCLs restorations) | 32 | 32 | 32 | 32 | 32 | 33
NCCLs restorations
  (A)-No evidence | 28 | 29 | 28 | 29 | 30 | 32
  (B)-Evidence | 1 | 1 | 1 | 1 | 2 | 1
  NCCLs restorations missing | 3 | 2 | 3 | 2 | 0 | 0
Statistical Analysis 1: Comparison: FBDC-SE (G1; Control Group) vs FBU-SE (G4) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC by Self-Etch mode (FBDC-SE; G1) and MM adhesives by SE mode (MM-SE; G4G6) result in similar (no significant differences) Gingival Bleeding performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.132, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Gingival Bleeding-USPHS comparison between G1 and G4G6 Arms performance from baseline to 24 month recall
Statistical Analysis 2: Comparison: FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs ADU-ER (G5); H0 - Bonding to NCCLs with FBDC by SE and enamel etching mode (FBDC-SE-EE; G2) and MM adhesives by Etch-and-Rinse mode (MM-ER; G3G5) result in similar (no significant differences) Gingival Bleeding performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.257, Wilcoxon (Mann-Whitney) — Applied for rows/categories No Evidence vs Evidence of Gingival Bleeding-USPHS comparison between G2 and G3G5 Arms performance from baseline to 24 month recall
Statistical Analysis 3: Comparison: FBDC-SE (G1; Control Group) vs FBDC-SE-EE (G2; Control Group) vs FBU-ER (G3) vs FBU-SE (G4) vs ADU-ER (G5) vs ADU-SE (G6); H0 - Bonding to NCCLs with FBDC (G1G2) or FBU (G3G4), DC adhesives, and ADU (G5G6) light-curing adhesive, with SE or SE-ER/ER modes result in similar (no significant differences) Gingival Bleeding performance at 24 month follow-up recall; Test type: Equivalence — An alpha value of 0.05 was considered; p = 0.918, Kruskal-Wallis — Applied for rows/categories No Evidence vs Evidence of Gingival Bleeding-USPHS comparison between G1G2 and G3G4 and G5G6 Arms performance from baseline to 24 month recall. P-value adjusted

ADVERSE EVENTS:
Time Frame: From baseline to 24th month recall.
Arm/Group | FBDC-SE (G1; Control Group) | FBDC-SE-EE (G2; Control Group) | FBU-ER (G3) | FBU-SE (G4) | ADU-ER (G5) | ADU-SE (G6)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-08-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT02698371/Prot_SAP_ICF_000.pdf